CLINICAL TRIAL: NCT03537404
Title: A Drug Interaction Study to Assess the Pharmacokinetics of Narlaprevir and Antiretroviral Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: Almedis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ05013019
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: hepatitis C; chronic; pharmacokinetics; HIV; coinfection; concomitant therapy
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome; Coinfection | interventions — narlaprevir; Ritonavir; Tenofovir; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment A (Part 1/ Part 2) (Active Comparator): Narlaprevir 200 mg once daily with Ritonavir 100 mg once daily for 5 days
  Interventions: Drug: Narlaprevir; Drug: Ritonavir
- Treatment B (Part 1) (Active Comparator): Tenofovir disoproxil fumarate 300 mg once daily for 5 days
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- Treatment B (Part 2) (Active Comparator): Raltegravir 400 mg twice daily for 5 days
  Interventions: Drug: Raltegravir
- Treatment C (Part 1) (Experimental): Narlaprevir 200 mg once daily coadministered with ritonavir 100 mg once daily and Tenofovir disoproxil fumarate 300 mg once daily for 5 days
  Interventions: Drug: Narlaprevir; Drug: Ritonavir; Drug: Tenofovir Disoproxil Fumarate
- Treatment C (Part 2) (Experimental): Narlaprevir 200 mg once daily coadministered with ritonavir 100 mg once daily and 400 mg raltegravir twice daily for 5 days
  Interventions: Drug: Narlaprevir; Drug: Ritonavir; Drug: Raltegravir

INTERVENTIONS:
Drug: Narlaprevir — 100 mg, film-coated tablets, taken as 200 mg per os daily
  Other Names: Arlansa
  Arms: Treatment A (Part 1/ Part 2); Treatment C (Part 1); Treatment C (Part 2)
Drug: Ritonavir — 100 mg, film-coated tablets, taken as 100 mg per os daily
  Other Names: Norvir
  Arms: Treatment A (Part 1/ Part 2); Treatment C (Part 1); Treatment C (Part 2)
Drug: Tenofovir Disoproxil Fumarate — 300 mg, film-coated tablets, taken as 300 mg per os daily
  Other Names: Tenofovir-TL; Viread
  Arms: Treatment B (Part 1); Treatment C (Part 1)
Drug: Raltegravir — 400 mg, film-coated tablets, taken as 400 mg per os daily
  Other Names: Isentress
  Arms: Treatment B (Part 2); Treatment C (Part 2)

SUMMARY:
The study purpose is to evaluate the potential for a pharmacokinetic drug-drug interaction, safety and tolerability when Narlaprevir, Ritonavir (used as a metabolic inhibitor) and Tenofovir disoproxil fumarate (part 1) and Narlaprevir, Ritonavir and Raltegravir (part 2) are administered in combination to healthy volunteers.

DETAILED DESCRIPTION:
The current study includes 2 parts, as the following drugs may be used concomitantly to treat hepatitis C virus (HCV)/HIV coinfection:

* Part 1 of the study is being conducted to evaluate the pharmacokinetic effect of coadministration of narlaprevir with ritonavir and tenofovir disoproxil fumarate.
* Part 2 of the study is being conducted to evaluate the pharmacokinetic effect of coadministration of narlaprevir/ritonavir and raltegravir.

Each part of the study is designed as a randomized 3-period crossover study and will assess if there is any effect of tenofovir disoproxil fumarate or raltegravir on the pharmacokinetics of narlaprevir and vice versa.

Subjects will be screened within 28 days before dosing in this multi-part study. All subjects eligible for protocol criteria will be randomized 1:1:1 to receive one of the following treatment sequences: A/B/C, or B/C/A, or C/A/B. Every subject will receive only one treatment (A or B or C) in one Period. Subjects will be confined to the study center throughout treatment in each period. Following completion of study procedures for each treatment period, subjects will be released from the clinic. After a 7-14 (maximum) days interval between dosing, subjects will return to start hospitalization for the next treatment period. Subjects will be discharged from the study upon completion of all study related procedures in Period 3. Phone call will be conducted after 5-7 days of follow-up period to assess safety data.

This drug interaction study is designed to investigate pharmacokinetic drug-drug interactions between Narlaprevir coadministered with Ritonavir and antiretroviral drugs (Tenofovir disoproxil fumarate and Raltegravir) for labeling and clinical dosing guidance purposes.

ELIGIBILITY:
Inclusion Criteria (the subject must meet all the criteria listed below for entry at baseline and at Days -1 and 1 before each treatment Period):

* Subjects must be willing to give written informed consent for the trial and able to adhere to dose and visit schedules.
* Subjects having a Body Mass Index (BMI) between 18,5 and 30 kg/m^2, inclusive.
* Subjects should diagnosed as "healthy": no pathology of the gastrointestinal tract, liver, kidneys, cardiovascular system, central nervous system (previously carried out by standard clinical and lab tests which did not reveal the presence of any diseases. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must not exceed the normal range; QT interval calculated by Bazett's formula (QTcB) for men should be ≤ 450 ms and ≤ 470 ms for women, the interval PR should be ≤ 200 ms).
* Vital sign measurements (taken after ~3 minutes in a supine or sitting position) must be within the following ranges:

  1. systolic blood pressure, 100 - 130 mm Hg;
  2. diastolic blood pressure, 60 -90 mm Hg;
  3. pulse rate, 60-80 bpm.
* Female subjects must be:

  1. postmenopausal (defined as 12 months with no menses; age > 40 years and with a follicle-stimulating hormone (FSH) level of >40 u/mL);
  2. surgically sterilized at least 3 months prior to baseline (e.g., documented hysterectomy or tubal ligation).
* Men must agree to use a medically accepted method of contraception (condom and spermicide) during the trial and for 3 months after stopping the medication.

Exclusion Criteria (the subject will be excluded from entry if any of the criteria listed below are met at baseline):

* Females with childbearing potential.
* Subjects who, in the opinion of the investigator, will not be able to participate optimally in the study.
* Positive results for hepatitis B surface antigen, hepatitis C antibodies or HIV, positive RW results.
* Allergic reactions in history.
* Intolerance to medication.
* Chronic disease of cardiovascular, bronchopulmonary, and/or neuroendocrine systems, gastrointestinal, liver, pancreas, kidney and/or blood disease.
* History or presence of impaired renal function, lactase deficiency, lactose intolerance, glucose-galactose malabsorption.
* History of urinary obstruction or difficulty in voiding.
* Gastrointestinal surgery in history (except of appendectomy).
* Acute infections less than 4 weeks before participation in the study.
* Subjects with a medical history of osteopenia and/or osteoporosis.
* Regular administration of any medicines less than 4 weeks before participation in the study.
* Administration of medicines with marked influence on hemodynamics, liver function et al (barbiturates, omeprazole, cimetidine et al) less than 30 days before participation in the study.
* Blood donation (450 ml or more of blood or plasma) less than 2 months before participation in the study.
* Intake of more than 10 units of alcohol in a week (1 unit of alcohol is equal to 0.5 L of beer, 200 mL of wine or 50 mL of spirits) or history of drug abuse or alcoholism.
* Smoking of more than 10 cigarettes or equivalent tobacco use per day.
* Participation in phase 1 clinical trial less than 3 months before participation in the study.
* Positive screen for drugs abuse and drugs use.
* Subjects with a medical history of psychiatric or personality disorders that in the opinion of the investigator and sponsor, affects the subject's ability to participate in the trial.
* Subjects who are part of the study staff personnel or family members of the study staff personnel.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-06-24 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (1):
- Clinic "Bessalar" JSC, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult volunteers were recruited for all Parts of the study in one clinical site (Bessalar clinic) in Moscow between April and June 2017. 36 subjects were randomized so that 18 subjects participated in each Part of the study (6 subjects in each treatment group of each Part).
Pre-assignment Details: Subjects were to be screened within 28 days before dosing in this multi-part study. Subjects were to be admitted to the study center the evening before the first dose for baseline assessments to confirm eligibility.
Groups:
- Part 1: All patients of Part 1 of the study were randomized in 1:1:1 ratio to receive one of the treatment sequences (A/B/C, B/C/A or C/A/B). Every subject received only one drug combination (A or B or C) in one treatment period. Each period was followed by 8 washout days. Treatments include:
  Narlaprevir (100 mg, film-coated tablets, taken as 200 mg per os once daily); Ritonavir (100 mg, film-coated tablets, taken as 100 mg per os once daily); Tenofovir Disoproxil Fumarate (300 mg, film-coated tablets, taken as 300 mg per os once daily) in different combinations assigned to the subjects in accordance with protocol considerations for Part 1 of the study.
- Part 2: All patients of Part 2 of the study were randomized in 1:1:1 ratio to receive one of the treatment sequences (A/B/C, B/C/A or C/A/B). Every subject received only one drug combination (A or B or C) in one treatment period. Each period was followed by 8 washout days. Treatments include:
  Narlaprevir (100 mg, film-coated tablets, taken as 200 mg per os once daily); Ritonavir (100 mg, film-coated tablets, taken as 100 mg per os once daily); Raltegravir (400 mg, film-coated tablets, taken as 400 mg per os once daily) in different combinations assigned to the subjects in accordance with protocol considerations for Part 2 of the study.
Period: First Intervention (A or B or C)
Arm/Group | Part 1 | Part 2
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: First Washout Period (8 Days)
Arm/Group | Part 1 | Part 2
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Second Intervention (A or B or C)
Arm/Group | Part 1 | Part 2
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Second Washout Period (8 Days)
Arm/Group | Part 1 | Part 2
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Third Intervention (A or B or C)
Arm/Group | Part 1 | Part 2
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 36 subjects randomized to study treatment and received at least one dose of study drug (Safety Population).
Groups:
- Sequence A/B/C: All participants of Part 1 or 2 of the study randomized in this group received treatment combinations (according to the protocol allocation) in the following sequence:
  Treatment period 1 - Treatment A Treatment period 2 - Treatment B Treatment period 3 - Treatment C
- Sequence B/C/A: All participants of Part 1 or 2 of the study randomized in this group received treatment combinations (according to the protocol allocation) in the following sequence:
  Treatment period 1 - Treatment B Treatment period 2 - Treatment C Treatment period 3 - Treatment A
- Sequence C/A/B: All participants of Part 1 or 2 of the study randomized in this group received treatment combinations (according to the protocol allocation) in the following sequence:
  Treatment period 1 - Treatment C Treatment period 2 - Treatment A Treatment period 3 - Treatment B
- Total: Total of all reporting groups
Arm/Group | Sequence A/B/C | Sequence B/C/A | Sequence C/A/B | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics analisys was performed separately for Part 1 and 2 of the study (18 subjects in each Part were randomized in 1:1:1 ratio for each treatment sequence - 6 participants in each).
  years
    Part 1: number analyzed (Participants) | 6 | 6 | 6 | 18
    Part 1 | 24.3 (1.75) | 38.3 (8.26) | 29.7 (1.86) | 30.8 (7.57)
    Part 2: number analyzed (Participants) | 6 | 6 | 6 | 18
    Part 2 | 24.3 (4.03) | 38.7 (4.59) | 29.5 (3.33) | 30.8 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics analisys was performed separately for Part 1 and 2 of the study (18 subjects in each Part were randomized in 1:1:1 ratio for each treatment sequence - 6 participants in each).
  Participants
    Part 1: number analyzed (Participants) | 6 | 6 | 6 | 18
    Part 1: Female | 0 | 0 | 0 | 0
    Part 1: Male | 6 | 6 | 6 | 18
    Part 2: number analyzed (Participants) | 6 | 6 | 6 | 18
    Part 2: Female | 0 | 0 | 0 | 0
    Part 2: Male | 6 | 6 | 6 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics analisys was performed separately for Part 1 and 2 of the study (18 subjects in each Part were randomized in 1:1:1 ratio for each treatment sequence - 6 participants in each).
  Participants
    Part 1: number analyzed (Participants) | 6 | 6 | 6 | 18
    Part 1: White | 6 | 6 | 5 | 17
    Part 1: Asian | 0 | 0 | 1 | 1
    Part 1: Black | 0 | 0 | 0 | 0
    Part 1: Other | 0 | 0 | 0 | 0
    Part 2: number analyzed (Participants) | 6 | 6 | 6 | 18
    Part 2: White | 6 | 5 | 6 | 17
    Part 2: Asian | 0 | 1 | 0 | 1
    Part 2: Black | 0 | 0 | 0 | 0
    Part 2: Other | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Calculated as weight(kg)/height(m^2) Population: Baseline characteristics analisys was performed separately for Part 1 and 2 of the study (18 subjects in each Part were randomized in 1:1:1 ratio for each treatment sequence - 6 participants in each).
  kg/m2
    Part 1: number analyzed (Participants) | 6 | 6 | 6 | 18
    Part 1 | 23.14 (1.287) | 24.73 (3.022) | 24.20 (3.134) | 24.02 (2.554)
    Part 2: number analyzed (Participants) | 6 | 6 | 6 | 18
    Part 2 | 24.26 (4.132) | 25.40 (2.732) | 25.63 (3.408) | 25.10 (3.319)

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Narlaprevir
Description: Maximum observed Concentration of Narlaprevir at Day 5 of treatment A and C of Part 1 or 2 of the study
Time Frame: Day 5 Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose on Day 5 of treatment A and C (Part 1/ Part 2)
Population: All subjects randomized to study treatment and received at least one dose of study drug.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/ml
Groups:
- Treatment A (Part 1); Treatment A (Part 2): Subjects in both Parts of the study recieved as Treatment A for 5 days (in respective treatment period):
  Narlaprevir (100 mg, film-coated tablets, taken as 200 mg per os once daily) and Ritonavir (100 mg, film-coated tablets, taken as 100 mg per os once daily).
- Treatment C (Part 1): Subjects recieved as Treatment C for 5 days (in respective treatment period):
  Narlaprevir (100 mg, film-coated tablets, taken as 200 mg per os once daily) coadministered with Ritonavir (100 mg, film-coated tablets, taken as 100 mg per os once daily) and Tenofovir Disoproxil Fumarate (300 mg, film-coated tablets, taken as 300 mg per os once daily).
- Treatment C (Part 2): Subjects recieved as Treatment C for 5 days (in respective treatment period):
  Narlaprevir (100 mg, film-coated tablets, taken as 200 mg per os once daily) coadministered with Ritonavir (100 mg, film-coated tablets, taken as 100 mg per os once daily and Raltegravir (400 mg, film-coated tablets, taken as 400 mg per os twice daily).
Arm/Group | Treatment A (Part 1) | Treatment C (Part 1) | Treatment A (Part 2) | Treatment C (Part 2)
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng/ml | 2130.2742 [1817.4088 to 2731.8348] | 2172.233 [1895.673 to 2726.557] | 2946.131 [2617.485 to 3799.642] | 2880.612 [2412.858 to 4121.871]
Statistical Analysis 1: Comparison: Treatment A (Part 1) vs Treatment C (Part 1); Test type: Other; Geometric Mean Ratio = 0.020, 90% CI 2-sided [-0.103 to 0.142] — Cmax parameters were logarithmically transformed
Statistical Analysis 2: Comparison: Treatment A (Part 2) vs Treatment C (Part 2); Test type: Other; Geometric Mean Ratio = -0.022, 90% CI 2-sided [-0.220 to 0.175] — Cmax parameters were logarithmically transformed

2. Primary Outcome: AUCtau of Narlaprevir
Description: Area Under the Concentration-time curve during a dosing interval τ at steady state of Narlaprevir at Day 5 of treatment A and C of Part 1/ Part 2 of the study
Time Frame: as for outcome 1
Population: All subjects randomized to study treatment and received at least one dose of study drug.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/ml
Arm/Group | Treatment A (Part 1) | Treatment C (Part 1) | Treatment A (Part 2) | Treatment C (Part 2)
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng*h/ml | 20504.31 [18265.63 to 24328.95] | 21366.2 [18664.1 to 26481.9] | 26199.19 [23136.15 to 33132.53] | 24458.48 [20738.76 to 33597.42]
Statistical Analysis 1: Comparison: Treatment A (Part 1) vs Treatment C (Part 1); Test type: Other; Geometric Mean Ratio = 0.041, 90% CI 2-sided [-0.075 to 0.157] — AUCtau parameters were logarithmically transformed
Statistical Analysis 2: Comparison: Treatment A (Part 2) vs Treatment C (Part 2); Test type: Other; Geometric Mean Ratio = -0.069, 90% CI 2-sided [-0.201 to 0.064] — AUCtau parameters were logarithmically transformed

3. Primary Outcome: Cmax of Tenofovir
Description: Maximum observed Concentration of Tenofovir at Day 5 of treatment B and C of Part 1 of the study
Time Frame: Day 5 Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 18 and 24 hrs post-dose on Day 5 of treatment B and C (Part 1)
Population: All subjects randomized to study treatment and received at least one dose of study drug.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/ml
Groups:
- Treatment B (Part 1): Subjects recieved as Treatment B for 5 days (in respective treatment period):
  Tenofovir Disoproxil Fumarate (300 mg, film-coated tablets, taken as 300 mg per os once daily).
Arm/Group | Treatment B (Part 1) | Treatment C (Part 1)
Number analyzed (Participants) | 18 | 18
ng/ml | 263.037 [233.126 to 313.318] | 344.796 [302.457 to 415.092]
Statistical Analysis 1: Comparison: Treatment B (Part 1) vs Treatment C (Part 1); Test type: Other; Geometric Mean Ratio = 0.271, 90% CI 2-sided [0.159 to 0.383] — Cmax parameters were logarithmically transformed

4. Primary Outcome: AUCtau of Tenofovir
Description: Area Under the Concentration-time curve during a dosing interval τ at steady state of Tenofovir at Day 5 of treatment B and C of Part 1 of the study
Time Frame: Day 5 Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 18 and 24 hrs post-dose on Day 5 of treatment B and C (Part 1)
Population: All subjects randomized to study treatment and received at least one dose of study drug.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/ml
Arm/Group | Treatment B (Part 1) | Treatment C (Part 1)
Number analyzed (Participants) | 18 | 18
ng*h/ml | 2599.95 [2325.72 to 3043.02] | 2799.72 [2536.67 to 3205.65]
Statistical Analysis 1: Comparison: Treatment B (Part 1) vs Treatment C (Part 1); Test type: Other; Geometric Mean Ratio = 0.074, 90% CI 2-sided [0.016 to 0.132] — AUCtau parameters were logarithmically transformed

5. Primary Outcome: Cmax of Raltegravir
Description: Maximum observed Concentration of Raltegravir at Day 5 of treatment B and C of Part 2 of the study
Time Frame: Day 5 Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12 hrs post-dose of Day 5 of treatment B and C (Part 2)
Population: All subjects randomized to study treatment and received at least one dose of study drug.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/ml
Groups:
- Treatment B (Part 2): Subjects recieved as Treatment B for 5 days (in respective treatment period):
  Raltegravir (400 mg, film-coated tablets, taken as 400 mg per os twice daily).
Arm/Group | Treatment B (Part 2) | Treatment C (Part 2)
Number analyzed (Participants) | 18 | 18
ng/ml | 830.204 [520.042 to 2758.109] | 715.726 [136.163 to 2396.130]
Statistical Analysis 1: Comparison: Treatment B (Part 2) vs Treatment C (Part 2); Test type: Other; Geometric Mean Ratio = -0.148, 90% CI 2-sided [-0.450 to 0.153] — Cmax parameters were logarithmically transformed

6. Primary Outcome: AUCtau of Raltegravir
Description: Area Under the Concentration-time curve during a dosing interval τ at steady state of Tenofovir at Day 5 of treatment B and C of Part 2 of the study
Time Frame: Day 5 Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12 hrs post-dose of Day 5 of treatment B and C (Part 2)
Population: All subjects randomized to study treatment and received at least one dose of study drug.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/ml
Arm/Group | Treatment B (Part 2) | Treatment C (Part 2)
Number analyzed (Participants) | 18 | 18
ng*h/ml | 2912.45 [1983.01 to 8451.44] | 2653.65 [1033.88 to 6964.58]
Statistical Analysis 1: Comparison: Treatment B (Part 2) vs Treatment C (Part 2); Test type: Other; Geometric Mean Ratio = -0.093, 90% CI 2-sided [-0.354 to 0.168] — AUCtau parameters were logarithmically transformed

7. Secondary Outcome: Number of Patients With Adverse Events
Time Frame: Up to 14 Days after the last dose of treatment in period 3 of each Part of the Study
Population: All subjects randomized to study treatment and received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Treatment A (Part 1); Treatment A (Part 2): Narlaprevir, 100 mg, film-coated tablets, taken as 200 mg per os daily in combination with Ritonavir, 100 mg, film-coated tablets, taken as 100 mg per os daily for 5 days
- Treatment B (Part 1): Tenofovir Disoproxil Fumarate, 300 mg, film-coated tablets, taken as 300 mg per os daily for 5 days
- Treatment C (Part 1): Narlaprevir, 100 mg, film-coated tablets, taken as 200 mg per os daily
  coadministered with
  Ritonavir, 100 mg, film-coated tablets, taken as 100 mg per os daily
  and
  Tenofovir Disoproxil Fumarate, 300 mg, film-coated tablets, taken as 300 mg per os daily for 5 days
- Treatment B (Part 2): Raltegravir, 400 mg, film-coated tablets, taken as 400 mg per os daily for 5 days
- Treatment C (Part 2): Narlaprevir, 100 mg, film-coated tablets, taken as 200 mg per os daily
  coadministered with
  Ritonavir, 100 mg, film-coated tablets, taken as 100 mg per os daily
  and
  Raltegravir, 400 mg, film-coated tablets, taken as 400 mg per os daily for 5 days
Arm/Group | Treatment A (Part 1) | Treatment B (Part 1) | Treatment C (Part 1) | Treatment A (Part 2) | Treatment B (Part 2) | Treatment C (Part 2)
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18
Participants | 1 | 0 | 4 | 0 | 0 | 1

8. Secondary Outcome: Number of Patients With Changes in Vital Signs
Description: There were no subjects with abnormal changes in vital signs
Time Frame: Up to 14 Days after the last dose of treatment in period 3 of each Part of the Study
Population: All subjects randomized to study treatment and received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A (Part 1) | Treatment B (Part 1) | Treatment C (Part 1) | Treatment A (Part 2) | Treatment B (Part 2) | Treatment C (Part 2)
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Patients With Abnormal Laboratory Values
Time Frame: Up to 14 Days after the last dose of treatment in period 3 of each Part of the Study
Population: All subjects randomized to study treatment and received at least one dose of study drug separately for each Patr of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A (Part 1) | Treatment B (Part 1) | Treatment C (Part 1)
Number analyzed (Participants) | 18 | 18 | 18
Participants
  Part 1 | 0 | 0 | 2
  Part 2 | 0 | 0 | 1

10. Secondary Outcome: Number of Patients With Abnormal ECG Changes
Description: There were no subjects with abnormal ECG changes during the study
Time Frame: Up to 14 Days after the last dose of treatment in period 3 of each Part of the Study
Population: All subjects randomized to study treatment and received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Treatment A (Part 1/Part 2): Narlaprevir, 100 mg, film-coated tablets, taken as 200 mg per os daily in combination with Ritonavir, 100 mg, film-coated tablets, taken as 100 mg per os daily for 5 days
- Treatment B (Part 1/Part 2): Part 1: Tenofovir Disoproxil Fumarate, 300 mg, film-coated tablets, taken as 300 mg per os daily for 5 days
  Part 2: Raltegravir, 400 mg, film-coated tablets, taken as 400 mg per os daily for 5 days
- Treatment C (Part 1/Part 2): Part 1: Narlaprevir, 100 mg, film-coated tablets, taken as 200 mg per os daily coadministered with Ritonavir, 100 mg, film-coated tablets, taken as 100 mg per os daily and Tenofovir Disoproxil Fumarate, 300 mg, film-coated tablets, taken as 300 mg per os daily for 5 days
  Part 2: Narlaprevir, 100 mg, film-coated tablets, taken as 200 mg per os daily coadministered with Ritonavir, 100 mg, film-coated tablets, taken as 100 mg per os daily and Raltegravir, 400 mg, film-coated tablets, taken as 400 mg per os daily for 5 days
Arm/Group | Treatment A (Part 1/Part 2) | Treatment B (Part 1/Part 2) | Treatment C (Part 1/Part 2)
Number analyzed (Participants) | 18 | 18 | 18
Participants
  Part 1 | 0 | 0 | 0
  Part 2 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 Days after the last dose of treatment in period 3 of each Part of the Study
Arm/Group | Treatment A (Part 1) | Treatment B (Part 1) | Treatment C (Part 1) | Treatment A (Part 2) | Treatment B (Part 2) | Treatment C (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 0/18 | 4/18 | 0/18 | 0/18 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (Part 1) (N=18) | Treatment B (Part 1) (N=18) | Treatment C (Part 1) (N=18) | Treatment A (Part 2) (N=18) | Treatment B (Part 2) (N=18) | Treatment C (Part 2) (N=18)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood Lactate Dehydrogenase Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public availiable only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03537404/Prot_SAP_000.pdf